CLINICAL TRIAL: NCT00158210
Title: Double-Blind Randomized Placebo Controlled Trial of Rivastigmine (Excelon) as a Potential Medication for Methamphetamine Abuse
Brief Title: Rivastigmine For Methamphetamine Dependent Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Dr Steven Shoptaw, UCLA Department of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18185-1; P50DA018185 (NIH); DPMCDA
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-09

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
Methamphetamine abuse has been steadily increasing over the past decade. Rivastigmine is a medication that may be helpful in treating methamphetamine dependence. The purpose of this study is to evaluate the effectiveness of rivastigmine in treating methamphetamine dependent individuals.

DETAILED DESCRIPTION:
Methamphetamine is a powerful stimulant that affects the central nervous system. Chronic methamphetamine use often leads to psychotic behavior. Rivastigmine is an acetylcholinesterase inhibitor that is currently approved to treat Alzheimer's-related dementia. The purpose of this study is to assess the efficacy of rivastigmine in treating methamphetamine dependent individuals.

Participants will be randomly assigned to either one of two dose levels of rivastigmine or placebo for 12 weeks. Participants will be assessed for cardiovascular, subjective, and reinforcing effects that are produced by methamphetamine. All participants will partake in contingency management sessions through Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English
* Not seeking treatment for methamphetamine dependence at study entry
* Meets DSM-IV criteria for methamphetamine abuse or dependence
* Smokes or intravenously uses methamphetamine
* Resting pulse between 50 and 90 beats per minute within 2 days prior to study entry
* Systolic blood pressure between 85 and 150 mmHg and diastolic blood pressure between 45 and 90 mmHg within 2 days prior to study entry
* Electrocardiogram demonstrating normal sinus rhythm, normal conduction, and no clinically significant arrhythmias
* Medical history and brief physical examination demonstrating no clinically significant contraindications for study participation

Exclusion Criteria:

* History or evidence of seizures or brain injury
* Previous adverse reaction to methamphetamine
* Neurological or psychiatric disorders (e.g., psychosis, bipolar illness, or major depression)
* Organic brain disease or dementia
* History of any psychiatric disorder that requires ongoing treatment or that would make study compliance difficult
* History of suicide attempts within the 3 months prior to study entry
* Heart disease or high blood pressure
* Family history of early cardiovascular morbidity or mortality
* Untreated or unstable medical illness, including neuroendocrine, autoimmune, liver, kidney, or active infectious disease
* HIV infected
* AIDS-defining illness
* Currently taking antiretroviral medication
* Pregnant or breastfeeding
* Unwilling to use an adequate method of contraception for the duration of the study
* History of respiratory illness (e.g., asthma, chronic coughing, and wheezing)
* Currently using alpha or beta agonists, theophylline, or other sympathomimetics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Methamphetamine abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Steve Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California - Los Angeles, Los Angeles, California, United States